CLINICAL TRIAL: NCT06158984
Title: Managing Dry Eye in Patients Using Glaucoma Drops
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: He Eye Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GLADQSLIP2023
Record Dates: First submitted 2023-02-07; First posted 2023-12-06 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Dry Eye
Keywords: Glaucoma; IPL; Diquafosol; Drug-induced Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes; Glaucoma | interventions — Intense Pulsed Light Therapy

STUDY DESIGN:
Intervention Model Description: Prospective, comparative pilot study
Who Masked: Investigator, Outcomes Assessor
Masking Description: Masked examiner for all clinical assessments will not involved in the data collection or group allocation procedure for this research. The investigator will not be aware of the two groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IPL group (Experimental): IPL group will use 2 sessions of IPL therapy, 15 days apart for the management of drug-induced dry eye in glaucoma patients.
  Interventions: Device: IPL
- Control group (No Intervention): The control group received no treatment

INTERVENTIONS:
Device: IPL — Intense pulse light (IPL) therapy is used for the treatment of drug-related dry eye in glaucoma patients.
  Other Names: Intense pulsed light
  Arms: IPL group

SUMMARY:
A single center randomized controlled trial on managing dry eye signs and symptoms in patients using anti-glaucoma eye drops.

DETAILED DESCRIPTION:
To compare the safety and efficacy of IPL therapy on drug-induced dry eye caused by long-term use of anti glaucoma drugs;

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Able and willing to comply with the treatment/follow-up schedule
* Bilateral signs and symptoms of dry eye disease

Exclusion Criteria:

* Participants with systemic immune-mediated illnesses, such as secondary Sjögren's syndrome or graft-versus-host disease
* Patients using topical medication(s) for the treatment of ocular disorders such as allergic conjunctivitis were excluded from the study.
* Previous ocular surgery or trauma
* 1-month history of blepharal and periorbital skin disease or allergies
* Severe dry eyes with corneal epithelial defect
* Limbic keratitis
* Pterygium
* Corneal neovascularization
* Breastfeeding
* Rheumatic immune systemic diseases
* Herpes zoster infection
* Pregnant women
* Allergic to fluorescein
* Contact lens wearers

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-10-03 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-02 (Actual)

PRIMARY OUTCOMES:
Non-invasive tear break-up time | Day-0 (baseline), 2-week, 4-weeks
  Changes in non-invasive initial tear film breaking time will be assessed using the Keratograph 5M (Oculus, Germany) topographer.
  Three sequentially readings will be captured, and the median value will be included in the final analysis. The median value will be recorded.

SECONDARY OUTCOMES:
Conjunctival hyperemia (RS score) | Day-0 (baseline), 2-week, 4-weeks
  Conjunctival hyperemia (RS score) will be assessed by keratograph image (Oculus, Germany) of 1156*873 pixels, redness score (RS) (accurate to 0.1 U) was displayed on the computer screen that ranged from 0.0 to 4.0.
Quality of meibum grade | Day-0 (baseline), 2-week, 4-weeks
  Meibum quality will be assessed under a slit-lamp:
  Five meibomian gland in the middle parts of the eyelid will be assessed using a scale of 0 to 3 for each gland (0 represented clear meibum; 1 represented cloudy meibum; 2 represented cloudy and granular meibum; and 3 represented thick, toothpaste like consistency meibum).
Expressibility of meibum grade | Day-0 (baseline), 2-week, 4-weeks
  Meibum expressibility will be assessed under a slit-lamp:
  Eight meibomian glands in the middle part will be evaluated on a scale of 0 to 3 (0 denoted that all glands expressible; 1 denoted that 3 to 4 glands expressible; 2 denoted those 1 to 2 glands expressible; and 3 denoted that no glands were expressible). The overall score was computed using the mean scores of these eight glands.
Conjunctivocorneal epithelial staining grade | Day-0 (baseline), 1-week, 2-weeks
  Conjunctivocorneal epithelial staining will be assessed under a slit-lamp:
  Conjunctivocorneal epithelial staining will be assess corneal and conjunctival epithelium damage. Double vital staining approach with two microliters of a preservative-free solution containing 1% lissamine green and 1% sodium fluorescein will be instilled in the conjunctival sac.
  The eye will be sectioned into three equal pieces (temporal conjunctiva, cornea, and nasal conjunctiva). Each region receives a maximum staining score of three points and a minimum of zero points. The combined scores from all three parts were then recorded on a scale ranging from 0 (normal) to 9 (severe).
Tear Film Lipid Layer | Day-0 (baseline), 2-week, 4-weeks
  Tear Film Lipid Layer interferometry will be assessed using DR-1 (Kowa, Nagoya, Japan).
OSDI Score | Day-0 (baseline), 2-week, 4-weeks
  Chinese translated, and validated OSDI (Allergan Inc, Irvine, USA) version will beused to assess and quantify DE symptom. The 12 items of the questionnaire can be tabulated into a score that ranges from 0 (no symptoms) to 100 (severe symptoms) points

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Eric Pazo, Study Chair — He Eye Hospital, Shenyang, China
Locations (1):
- He Eye Hospital, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang H, Qi Y, Chen J, Qin G, Xu L, He W, Yu S, Che H, Pazo EE. Management of Glaucoma-Related Dry Eye Disease with Intense Pulsed Light: A Randomized Control Study. Clin Ophthalmol. 2024 Jul 15;18:2061-2072. doi: 10.2147/OPTH.S471426. eCollection 2024. PMID 39055379